CLINICAL TRIAL: NCT04160598
Title: Effect of Intravenous Magnesium on Post-spinal Fentanyl Induced Pruritus Incidence; A Prospective Randomized Controlled Study
Brief Title: Effect of Intravenous Magnesium on Post-spinal Fentanyl Induced Pruritus Incidence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R.19.09.628.R1.R2
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Magnesium Infusion in Post-spinal Opioid Pruritis
Keywords: Neuraxial opioids, post-operative itching, intrathecal Fentanyl pruritus, Spinal anesthesia
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): bolus 50 ml nacl 0.9% at the end of surgery over 20 minutes 5ml/minute infusion rate.
  Interventions: Drug: IV infusion; Drug: intrathecal fentanyl
- IV Mg ++ group (Experimental): continuous IV infusion pump of Magnesium 10mg/kg in 50 ml Nacl0.9% over 20 minutes at end of surgery 5ml/minute infusion rate.
  Interventions: Drug: IV infusion; Drug: intrathecal fentanyl

INTERVENTIONS:
Drug: IV infusion — Control group (Placebo Group): bolus 50 ml Nacl 0.9% at the end of surgery over 20 minutes 5ml/minute infusion rate.
Drug: intrathecal fentanyl — 10-15mg hyperbaric bupivacaine and 30µg fentanyl intrathecally injected

SUMMARY:
Introduction: Adding opioids to local anesthetic solutions leads to enhanced anesthesia and provide postoperative analgesia. Intrathecaly injected opioids have some side effects, though. One of them is pruritus. Objective: We designed a randomized, double-blinded, placebo-controlled study to evaluate prophylactic impact of continuous IV Magnesium 10mg/kg over 30 minutes on intrathecal fentanyl-induced pruritus start at the end of the operation.

Methods: ASA I-II Patient's candidate for orthopedic operations under spinal anesthesia (10-15mg hyperbaric bupivacaine and 25 µg fentanyl intrathecal) and will be divided randomly into two groups:

Control group (Placebo group): bolus 100 ml nacl 0.9% at end of surgery Study group (Mg ++ group): (continuous IV Magnesium 10mg/kg in 100 ml Nacl0.9% over 30 minutes at end of surgery).

Study outcome:

1. Hemodynamics: Systolic blood pressure, Mean arterial blood pressure, pulse rate, O2 saturation will be recorded in 5 min,10 min,30 min,60 min and every one hour till 6 hours after the operation.
2. Pruritus Patients were asked about existence (present=1,no=0), severity (mild=1, modret=2, sever =3) and site of pruritus (Face(trigeminal) =1, neuroaxial(dermatome)=2), 1,2,4, and 6 hours after operation. Incidence of pruritus total group incidence %.
3. The incidence of PONV.

DETAILED DESCRIPTION:
Study hypothesis Intravenous Magnesium would reduce and improve post-spinal fentanyl pruritus incidence outcome relaying up on the fact that Magnesium ions block the neuroaxial NMDA receptor which are involved in histamine-induced expansion of mechanical receptive field area, a neural event possibly involved in the development of pruritis. (36) Aim of the work To introduce Magnesium sulphate as cheap effective alternative for prevention and management of post-spinal opioid pruritis.

Methods This prospective randomized double blinded controlled study will be carried out in Mansoura faculty of medicine in Mansoura University hospital on cases subjected to LL orthopedic operations under spinal anesthesia utilizing bupivacaine plus adjuvant fentanyl which is documented to have high incidence of postspinal pruritus.

Patients: ASA I-II, of both genders, aged 20-70 years old Patient's candidate for LL orthopedic operations under spinal anesthesia. Total patient number of 144, will be enrolled into two groups 72 patients each, all patients will be anesthetized intrathecaly using10-15mg hyperbaric bupivacaine and 30 µg fentanyl and will be subdivided randomly into two groups:

Control group (Placebo Group): bolus 50 ml Nacl 0.9% at the end of surgery over 20 minutes 5ml/minute infusion rate.

Study group (MG++ Group): continuous IV infusion pump of Magnesium 10mg/kg in 50 ml Nacl0.9% over 20 minutes at end of surgery 5ml/minute infusion rate.

Randomization and blindness; the study drugs were prepared in 50 ml saline syringe according to the study randomization envelop method by an anesthesiologist who did not participate in the care and evaluation of the patients. The investigator and the patients were not aware of the drug they received.

Study outcomes (were assessed by the same clinician who cared for the patients in the perioperative and postoperative periods.)

1. Demographic data Age weight, length, BMI, operative type and operative time.
2. Hemodynamics:

   Systolic blood pressure, mean arterial blood pressure, heart rate, O2 saturation will be recorded basal, 10 min, 30 min, 60 min and every one hour till 6 hours after operation then every 6 h for the 1st 12 h after surgery.
3. Pruritus Primary outcome =Incidence of pruritus in each group incidence %. Includes 3 items 1. Existence (present=1, no=0), 2. Severity (mild=1, modret=2, sever =3) 3. Site of pruritus (Face (trigeminal) =1, neuraxial (dermatome) =2) during the 1st 6 hours after spinal fentanyl injection.
4. PO 1st 24 h Magnesium dose.
5. PO 1st 24 h Naloxone.
6. The incidence of PO vomiting% in each group. -Exclusion Criteria: BMI>35, Patient refusal, Hypersensitivity to amide local anesthetics, Fentanyl opioids, Magnesium and naloxone. Patients with coagulopathy, hepatic failure, LBBB and trifacicular block, General contraindications to spinal anesthesia, surgeon total refusal, Cardiac, hepatic, renal or respiratory failure, Difficult communication with the patient (psychological or deafness).

Side effects Management:

1. Residual Sever pruritus after the 1st magnesium bolus will be controlled 1st by 2 second postoperative 10mg/kg dose of magnesium bolus IV if not controlled within one hour Naloxone bolus dose of 0.4 mg then if pruritus attack not controlled another 0.4 mg naloxone in 100ml normal saline iv infusion over the next 1hour during the postoperative 12 hours.
2. Moderate Abdominal Pain: VAS >4 during surgical manipulation is unaccepted and managed soon using multimodal analgesia regimen including; ketorolac slow injection in an IV bolus of 0.5mg/kg if general anesthesia needed to control pain case will be excluded from the study.
3. Nausea & Vomiting: treated by metoclopramide 10 mg, if resistant IV bolus ondansetron 4mg, with treatment of hypotension if present.
4. Hypotension (mean arterial blood pressure (MAP) less than 65 mmHg, will be managed by using ephedrine bolus doses of 6mg, fluids and blood transfusion according to events and requirements.
5. Bradycardia (HR less than 60 b/m.) will be managed by atropine bolus of 0.5 mg.
6. Desaturation (SaO2< 90%) will be managed by increase oxygen face mask flow up to 10 L/sec. and dealing with the airway according to the situation targeting a patient airway with breathing comfort and O2saturation>94% In case of any respiratory depression, emergency airway equipment's and drugs for resuscitation for airway management and ventilation were kept ready.

   * Sample size calculation Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 15.0.5 for windows (2017) using the results published by [S.S. Jahanbakhsh and S. Bazyar. Study on prophylactic impact of ondansetron IV on intrathecal fentanyl-induced pruritus. British Journal of Anesthesia 108 (S2): ii387-ii437 (2012) doi:10.1093/bja/aer489] (37) With the incidence of post-operative opioid induced pruritis after spinal anesthesia as the primary outcome. Patients will be allocated into two groups: control group (placebo Group) and the study group (MG++ Group). Jahanbakhsh 2012 resulted in post-spinal fentanyl induced pruritus incidence of 34% ondansetron group versus 60% in the placebo group. The null hypothesis is assumed to be the absence of difference between both treatment modalities. A sample of 65 patients is in each group needed to achieve 80% power (1-β or the probability of rejecting the null hypothesis when it is false) to detect a difference between the group proportions of 26% using two-sided Fisher's exact test with a significance level of 0.05(α or the probability of rejecting the null hypothesis when it is true). The expected number of dropouts is 7 patients in each group so 72 patients will be enrolled into each group with a total study sample size number of 144 patients.

Statistical analysis IBM's SPSS Statistics (Statistical Package for the Social Sciences) for Windows (version 25) will be used for statistical analysis of the collected data. Shapiro-Wilk test will be used to check the normality of the data distribution. Normally distributed continuous variables will be expressed as mean ± SD while categorical variables and the abnormally distributed continuous ones will be expressed as median and inter-quartile range or number and percentage (as appropriate). Student t-test and Mann-Whitney will be used for normally and abnormally distributed continuous data respectively. Chi-square tests will be used for categorical data using the crosstabs function. All tests will be conducted with a 95% confidence interval. If needed, bivariate correlations will be assessed using Pearson's or Spearman's correlation coefficient depending on the nature of data. P (probability) value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II Both genders Aged 20-70 years old Patient's candidate for LL orthopedic operations under spinal anesthesia

Exclusion Criteria:

BMI>35 Patient refusal Hypersensitivity to amide local anesthetics Fentanyl opioids Magnesium and naloxone. Patients with LBBB and trifacicular block General contraindications to spinal anesthesia surgeon total refusal Cardiac, hepatic, renal or respiratory failure Difficult communication with the patient (psychological or deafness).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pruritus in each group incidence %. | during the 1st 6 hours after spinal fentanyl injection.
  Existence,Severity, Site of pruritus (Face (trigeminal) =1, neuraxial (dermatome) =2)

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ghanem, Study Chair — Mansoura Faculty of Medicine-Mansoura University
Locations (1):
- Anesthesia department,Faculty of medicine, Mansoura univerisety, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No